CLINICAL TRIAL: NCT03053518
Title: Validation of Machine Learning Based Personalized Nutrition Algorithm to Reduce Postprandial Glycemic Excursions Among North American Individuals With Newly Diagnosed Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol Withdrawn
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-01059
Record Dates: First submitted 2017-02-02; First posted 2017-02-15 (Actual); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-08

CONDITIONS: Type2 Diabetes
Keywords: Type 2 Diabetes; Hyperglycemia; Personal Nutrition Project
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Investigators will recruit approximately 5 cohorts of 4 participants each for the sample size of 20 participants. A new cohort will be randomized approximately every 4 weeks. The maximum number of study participants at any point in the study will be 10.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Life Style (Active Comparator)
  Interventions: Behavioral: LifeStyle
- Life Style + Metformin (Experimental)
  Interventions: Device: Abbott Freestyle Libre Pro; Behavioral: LifeStyle

INTERVENTIONS:
Device: Abbott Freestyle Libre Pro — A professional, blinded, continuous glucose monitoring device will be inserted on the back of the upper arm to measure interstitial glucose every 5 min for 4 times / day.
  Other Names: Abbott
  Arms: Life Style + Metformin
Behavioral: LifeStyle — Isocaloric diets (breakfast, lunch, dinner, and 2 snacks), which will be prepared and delivered daily, including 2 days each of low, moderate, and high glycemic load (GL) foods.

SUMMARY:
This is an initial validation study of the Personal Nutrition Project (PNP) algorithm in a North American population with recently diagnosed Type 2 Diabetes (T2D). This is a 2-stage, single-group feeding study in 20 individuals, including 10 participants managed with lifestyle alone, and 10 managed with lifestyle plus metformin.

DETAILED DESCRIPTION:
The PNP algorithm, which uses a machine learning algorithm to predict postprandial glycemic, may be efficacious for generating tailored dietary advice to moderate the participant's glycemic response to food.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years to <70 years
* Diagnosed with T2DM within 2 years with an HbA1c<7%
* Diabetes management by metformin or lifestyle intervention
* Fasting C-peptide ≥ 0.5 mg/mL (0.17 nmol/L) (to exclude those for whom hyperglycemic exposure is driven by β-cell failure rather than dietary behaviors, as well as those requiring escalation of the medication regime)
* Ownership a smart phone and are willing to use it to monitor multiple factors influencing glycemic response to glycemia (e.g., sleep, physical activity, diet, stress, medication, and hunger)

Exclusion Criteria:

* are unable or unwilling to provide informed consent;
* are unable to participate meaningfully in an intervention that involves self-monitoring using software available in English (e.g., due to uncorrected sight impairment, illiterate, non-English-speaking, dementia);
* are pregnant, are currently trying to become pregnant, or who become pregnant during the study
* are institutionalized (e.g., in a nursing home or personal care facility, or those who are incarcerated and have limited control over self-management)
* have had or are planning to have bariatric surgery during the study
* have a history of heart disease, kidney disease, or retinopathy (to rule-out those with long-standing, undiagnosed T2D)
* those with an active infection requiring antibiotics in the last 3 months or who develop an active infection requiring antibiotics during the study;
* those who use acetaminophen and are unwilling or unable to discontinue its use during the study (acetaminophen affects CGM accuracy)39
* immunosuppressive drugs within three months prior to participation and
* Chronically active inflammatory or neoplastic disease in the three years prior to enrollment.
* Patients with known food allergy.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sevick, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Life Style + Metformin
Started | 22
Completed | 12
Not Completed | 10
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Ineligible | 5

BASELINE CHARACTERISTICS:
Arm/Group | Life Style + Metformin
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Observed Incremental Area Under the Curve (iAUCobs)
Description: Observed incremental area under the curve (iAUCobs) at 2 hours following each meal and snack will be evaluated via CGM using the Abbott Freestyle Libre Pro, which captures interstitial glucose every 5 minutes. A sensor is inserted into the participant's upper arm. Participants will be blinded to glycemia tracings.
Time Frame: 2 Hours
Population: There is not enough usable data collected to analyze primary outcome measure due to low adherence to the study.
Arm/Group | Life Style + Metformin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Life Style + Metformin
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT03053518/Prot_000.pdf